CLINICAL TRIAL: NCT05362695
Title: A Phase 1 Placebo-controlled Study of the Safety and Tolerability of Rectally Administered, Multiple-ascending Doses of IW-3300 in Healthy Subjects
Brief Title: A Study of Multiple-ascending Doses of IW-3300 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: C3300-102
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator and all other clinical research unit staff, sponsor study personnel, and the participant will remain blinded to individual participant treatment assignments throughout the study. Treatment assignments of individual participants will only be unblinded to a sponsor representative for regulatory reporting purposes or if warranted by emerging safety or tolerability issues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: 100 μg IW-3300 (Experimental): 100 μg dose of active drug (IW-3300) once daily for 7 days
  Interventions: Drug: IW-3300
- Cohort 1: Placebo (Placebo Comparator): matching placebo once daily for 7 days
  Interventions: Drug: Placebo
- Cohort 2: 300 μg IW-3300 (Experimental): 300 μg dose of active drug (IW-3300) once daily for 7 days
  Interventions: Drug: IW-3300
- Cohort 2: Placebo (Placebo Comparator): matching placebo once daily for 7 days
  Interventions: Drug: Placebo
- Cohort 3 (optional): Dose 3 (Experimental): Active drug (IW-3300) once daily for 7 days
  Interventions: Drug: IW-3300
- Cohort 3 (optional): Placebo (Placebo Comparator): Matching placebo once daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IW-3300 — A dose of IW-3300 administered rectally (as a low-volume [20 mL] enema).
  Arms: Cohort 1: 100 μg IW-3300; Cohort 2: 300 μg IW-3300; Cohort 3 (optional): Dose 3
Drug: Placebo — A dose of placebo administered rectally (as a low-volume [20 mL] enema).
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3 (optional): Placebo

SUMMARY:
This clinical study is designed as a multiple-ascending-dose, safety and tolerability study with IW-3300. The study drug will be administered as a low-volume [20 mL] enema. Study participants will be randomized in a 2:1 ratio to receive IW-3300 or placebo. Up to 3 different doses of IW-3300 will be studied. Safety reviews will be conducted before proceeding to each higher dose.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, randomized, double-blind, placebo-controlled, multiple-ascending-dose study of IW-3300 administered rectally, once-daily, for 7 days as a low-volume enema in healthy adult participants. This study will assess the effect of IW-3300 on safety and tolerability.

The study includes up to 4 treatments: placebo and up to 3 dose levels of IW-3300 which will be determined after safety reviews of previous cohorts.

The 9 participants within each cohort will be randomized to receive IW-3300 (6 subjects) or placebo (3 participants), administered rectally (as a low-volume [20 mL] enema). Participants in each dosing cohort will progress through 3 study periods: (1) Screening Period, (2) Clinic Period, and (3) Follow-up Period. Treatment duration will be 7 days; participants will be followed in the Phase 1 clinical research unit (CRU) for the duration of dosing, until at least 24 hours after the last dose of study drug and contacted by phone for follow-up approximately 2 weeks after the last dose. Total participant participation will be 29 to 57 days, including the Screening, Clinic, and Follow-up Periods.

ELIGIBILITY:
Inclusion Criteria:

* Males and female subjects of non-childbearing potential
* Ages 18 to 60 years
* Medically healthy with no clinically significant findings during medical evaluation including physical examination, 12-lead electrocardiogram (ECG), and clinical laboratory tests.
* Body mass index (BMI) within the range 18.5 to 35.0 kg/m^2 (inclusive) at the Screening Visit.
* Male subjects and female partners are willing to use double-barrier method of contraception during the study.

Exclusion Criteria:

* Evidence or history of clinically significant acute or chronic disease, or clinically significant illness within 30 days of the Screening Visit.
* History of clinically significant hypersensitivity or allergies to any of the inactive ingredients contained in the active or placebo drug products.
* History of any condition that would interfere with their ability to receive an enema, or has had difficulty receiving an enema in the past.
* Recent history of anal fissure, anal abscess, complicated hemorrhoids, or presence or history of inflammatory bowel disease.
* Abnormal laboratory tests or clinically significant findings on safety tests conducted at the Screening Visit or at Check-in.
* Positive serology for human immunodeficiency virus (HIV) 1, HIV 2, or hepatitis B surface antigen (HBsAg), or positive for anti-HIV 1, anti-HIV 2, or anti hepatitis C virus (HCV) antibodies at the Screening Visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ironwood Study Chair, Study Director — Ironwood Pharmaceuticals
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to include up to 3 cohorts with 9 participants per cohort. Within each cohort, participants were randomized to receive a single dose of IW-3300 (6 participants) or placebo (3 participants). Doses to be evaluated were 100 and 300 μg. An optional 3rd cohort was planned to test an IW-3300 dose of >100 μg but <300 μg. Based on a blinded review of safety and tolerability data from Cohorts 1 and 2, the Dose Escalation Committee decided not to enroll the optional 3rd Cohort.
Pre-assignment Details: As pre-specified by the statistical analysis plan, for the analyses reported herein, data from the 3 participants dosed with placebo in each of the 2 cohorts were pooled into a single placebo group (N=6).
Groups:
- Placebo: A dose of placebo administered rectally (as a low-volume [20 mL] enema) once daily for 7 days
- 100 μg IW-3300: A 100 μg dose of IW-3300 administered rectally (as a low-volume [20 mL] enema) once daily for 7 days
- 300 μg IW-3300: A 300 μg dose of IW-3300 administered rectally (as a low-volume [20 mL] enema) once daily for 7 days
Period: Overall Study
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (9.52) | 47.8 (13.50) | 49.0 (9.30) | 44.8 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 5
  Male | 6 | 5 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 4 | 6 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 5 | 11
  Black or African American | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a treatment-emergent AE (TEAE) if the AE started after initial study drug administration and within 1 day of the last dose of study drug.
Time Frame: From first dose of study drug through 24 hours post-Day 1 dose
Population: Safety Analysis Set (all participants who received any amount of study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300
Number analyzed (Participants) | 6 | 6 | 6
Participants | 3 | 3 | 2

2. Primary Outcome: Number of Participants With Serious TEAEs
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is lifethreatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; or other situations such as important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. An SAE was considered a treatment-emergent SAE (serious TEAE) if the SAE started after initial study drug administration and within 1 day of the last dose of study drug.
Time Frame: From first dose of study drug through 24 hours post-Day 1 dose
Population: Safety Analysis Set (all participants who received any amount of study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 24 hours post-Day 1 dose
Description: An AE was considered a treatment-emergent AE (TEAE) if the AE started after initial study drug administration and within 1 day of the last dose of study drug.
Arm/Group | Placebo | 100 μg IW-3300 | 300 μg IW-3300
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | 100 μg IW-3300 (N=6) | 300 μg IW-3300 (N=6)
Corneal irritation (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT05362695/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT05362695/SAP_001.pdf